CLINICAL TRIAL: NCT03147599
Title: Mebeverine For Daytime And Nocturnal Incontinence and After Orthotopic W-Ileal Neobladders - Assessment Of Efficacy And Quality Of Life Effect Within 1 Year Post-Surgery: A Randomized Controlled Study
Brief Title: Mebeverine For 1st Year Daytime And Nocturnal Incontinence After Orthotopic W-Ileal Neobladders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R/17.02.32
Record Dates: First submitted 2017-03-15; First posted 2017-05-10 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2017-05

CONDITIONS: Oncology; Incontinence; Incontinence, Daytime Urinary; Incontinence, Nighttime Urinary; Bladder Cancer; Orthotopic Neobladder
Keywords: Mebeverine; Incontinence; Orthotopic Neobladder
MeSH Terms: conditions — Neoplasms; Diurnal Enuresis; Nocturnal Enuresis; Urinary Bladder Neoplasms | interventions — mebeverine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mebeverine (Active Comparator): Coloverin (Mebeverine hydrochloride 135 mg)
  Interventions: Drug: Coloverin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coloverin — Mebeverine hydrochloride 135 mg
  Other Names: Mebeverine hydrochloride
  Arms: Mebeverine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized controlled trial to assess clinically the efficacy of the selective ileum spasmolytic mebeverine on daytime incontinence and nocturnal enuresis of orthotopic w-ileal neobladders and quality of life effect within 1 year post-surgery.

DETAILED DESCRIPTION:
In appropriately selected patients an orthotopic neobladder (ONB) permits the elimination of an external stoma and preservation of body image without compromising cancer control after radical cystectomy. Voiding dysfunction (VD) following ONB can be divided into failure to empty bladder or failure to store urine. Failure to empty bladder by angulation of urethra is the most common cause. Failure to store urine can occur during daytime, night-time or both. VD that persists beyond 6 to 12 months warrants urodynamics evaluation to determine the cause and suggest plane of therapy. Voiding dysfunction has a detrimental impact on quality of life.

Among the various bowel segments studied, the ileum is ideal for ONB creation. A spherical reservoir, reconfigured from a de-tubularized ileal segment, offers the most desirable attributes like, adequate capacity, low intraluminal pressure, and good compliance. The patient of ONB reported 4-25% rate of clean intermittent self-catheterisation (CISC) for incomplete emptying. Daytime incontinence was present in 13% of patients. The rate of nocturnal incontinence is usually higher in the range of 15-40% in recent metanalysis. The success of ONB rely on detubularization of intestinal segment, sufficient capacity and proper configuration and position in the pelvis. Adequate capacity is achieved by using sufficient length, folding, and creation an ellipsoid or spherical configuration. The ONB should hold approximately 500 cc of urine at low pressure (at < 15 cm H2O), empty completely (< 100 cc urine), four to five times daily and allow the patient to sleep without awakening, while maintain normal body image

loss of the vesico-urethral reflex 'guarding reflex' in which increased urethral sphincter tone parallel to bladder distension, decreased patient vigilance during sleep resulting in reduced muscle tone and urethral closing pressure, decreased sensitivity of the membranous urethra after radical cystectomy, involuntary high-amplitude contractions of the reservoir secondary to bowel peristalsis and shifting of free water from the reservoir wall into the hyperosmolar urine are the main factor causing global and nocturnal polyuria in patient with ONB. Final, there is also evidence suggesting an increase in bowel activity during sleep. Maximum urethral closing pressure (MUCP) is the primary component responsible for daytime continence in patients with an ONB. However, Koraitim et al. suggest that nocturnal incontinence depends on three reservoir parameters: maximal contraction amplitude, baseline reservoir pressure at mid capacity, and MUCP.

Mebeverine is a derivative of reserpine, which has relatively specific effects on smooth muscle cells without atropine-like side effects in humans. It directly blocks voltage-operated sodium channels and inhibits intracellular calcium accumulation. It is three times more potent than papaverine in inhibiting the peristaltic reflex of the ileum.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 years or older
2. ONB within 1 year post-surgery.

Exclusion Criteria:

1. Upper urinary tract deterioration
2. Uncontrolled diabetes mellitus
3. Evident local or pelvic recurrence
4. Adjuvant chemotherapy
5. Chronic retention
6. Pouch stones
7. Urethral stricture or urethro-ileal maldirection
8. Sensitivity to Mebeverine
9. Untreated chronic constipation
10. Active symptomatic urinary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of mebeverine on daytime and nocturnal incontinence by assessing continence status measured by standardized continence questionnaire | 10 months
  Outcome Measure by standardized continence questionnaire

SECONDARY OUTCOMES:
Effect of mebeverine on patient quality of life by assessing patient quality of life measured by quality of life questionnaire | 10 months
  Outcome Measure by quality of life questionnaire
Effect of mebeverine on orthotopic w-ileal neobladders urodynamics by assessing simple urodynamic parameter | 10 months
  Outcome Measure by pressure change measurement in centimetre of water.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abol-Enein, MD, Study Chair — Urology and Nephrology Center; Ahmed Mosbah, MD, Study Director — Urology and Nephrology Center; Ahmed Elhussein, MBBCH, Principal Investigator — Urology and Nephrology Center; Ahmed Elkarta, MBBCH, Principal Investigator — Urology and Nephrology Center; Mohamed Soltan, MBBCH, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Hassan Abol-Enein, MD, Phd (Study Chair)